## <u>Randomized Trial to Test the Effect of Rivaroxaban or Apixaban on Menstrual Blood</u> <u>Loss in WomEn (RAMBLE)</u>

## NCT02829957

The primary comparison is the frequency of study-defined abnormal uterine bleeding between women treated with apixaban, versus women treated with rivaroxaban. The plan was to compare these frequencies using 95% confidence intervals for the difference in proportions.